CLINICAL TRIAL: NCT03426306
Title: A Novel Lung Function Imaging Modality As a Preoperative Evaluation Tool (LIME)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-2216.cc
Record Dates: First submitted 2018-02-01; First posted 2018-02-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
Keywords: 4-Dimensional Computed Tomography
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 4DCT-ventilation (Experimental): The patient will undergo 4DCT imaging. The 4DCT imaging data along with image processing techniques will be used to generate a 4DCT-ventilation map. All surgical decisions will be based on the current standard of care imaging (VQ scans) and not on the 4DCT imaging results.
  Interventions: Diagnostic Test: 4DCT-Ventilation

INTERVENTIONS:
Diagnostic Test: 4DCT-Ventilation — 4DCT-ventilation is an imaging modality that provides superior image quality, reduced cost, and a faster imaging procedure compared to nuclear medicine VQ scans.

SUMMARY:
To evaluate the correlation between pre-surgical 4DCT-ventilation imaging and post-surgical lung function.

DETAILED DESCRIPTION:
To evaluate the correlation between pre-surgical 4-Dimensional Computed Tomography-ventilation (4DCT-ventilation) imaging and post-surgical lung function. To determine whether 4DCT-ventilation is a better predictor of post-surgical lung function than nuclear medicine imaging using pulmonary function tests (PFTs). To determine whether 4DCT-ventilation is a better predictor of post-surgical lung function than nuclear medicine imaging using quality of life (QOL) questionnaires. Evaluate cost-effectiveness of using 4DCT-ventialtion and VQ scans for pre-surgical assessment. To use longitudinal (pre and post-surgical) 4DCT-ventilation imaging to derive novel post-surgical prediction formulas.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all required (non-optional) study procedures and be available for the duration of the study.
3. Be a male or female aged 18 to 100.
4. Patient with lung cancer (presumed or biopsy proven) currently undergoing or having undergone evaluation for resection.
5. Lung function assessment required for pre-surgical evaluation at the discretion of the cardiothoracic surgeon.
6. Life expectancy greater than 3 months.

Exclusion Criteria:

1. Patients getting a planned wedge resection as the only thoracic resectional procedure.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Pre-Surgical Imaging and Post-Surgical Lung Function | Baseline visit to follow up visit, up to 9 months.
  Measure the correlation between pre-surgical 4-Dimensional Computed Tomography-ventilation (4DCT) imaging and post surgical lung function using a Percent Predicted Post-Operative Pulmonary Function Test (%PPO PFT).

SECONDARY OUTCOMES:
Ability of %PPO PFTs | Start of study to end of study, up to 2 years
  Use %PPO PFTs to determine if 4DCT-ventilation is a better predictor of post surgical lung function than nuclear medicine imaging
Quality of Life (QOL) | Start of study to end of study, up to 2 years
  Use QOL questionnaires to determine if 4DCT-ventilation is a better predictor of post surgical lung function than nuclear medicine imaging.
Cost-Effectiveness | Start of study to end of study, up to 2 years
  Determine the cost-effectiveness of 4DCT-ventialtion and VQ scans for pre-surgical assessment using Receiver Operator Characteristic (ROC) analysis.
Longitudinal Imaging Changes | Start of study to end of study, up to 2 years
  Derive novel post-surgical prediction formulas using longitudinal 4DCT-ventilation imaging

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Jones, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - UCHealth Memorial Hospital, Colorado Springs, Colorado

IPD SHARING:
Plan to Share IPD: No